CLINICAL TRIAL: NCT04823091
Title: Safety and Efficacy of Anti-CD7 CAR-Engineered T Cells for Relapsed/Refractory T Lymphoid Malignancies: a Single-center, Open-label, Non-randomized, Single-arm Clinical Study
Brief Title: Anti-CD7 CAR-Engineered T Cells for T Lymphoid Malignancies Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Beijing GoBroad Hospital Management Co.,Ltd (Unknown); Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR7-T-cells
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: T-Cell Lymphocytic Leukemia; T-Cell Chronic Lymphocytic Leukemia; T Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, T-Cell; Leukemia, Prolymphocytic, T-Cell; Lymphoma, T-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cyclophosphamide + anti-CD7 CAR-T Cells (Experimental): Patients will received lymphodepletion with fludarabine (30 mg/kg) and cyclophosphamide (250 mg/kg) on day -5, -4, and -3, followed by the infusion of CAR7-T cells with the dose of 1×10^6/kg and 2×10^6/kg (with an allowance of ±20%). If no dose-limited toxicity (DLT) emerges in the group, then the subsequent higher dose will be used in the next group. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level. The maximum dose could be extended.
  Interventions: Drug: Fludarabine + Cyclophosphamide + CAR7-T Cells

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide + CAR7-T Cells — fludarabine 30 mg/kg on day -5, -4, and -3; cyclophosphamide 250 mg/kg on day -5, -4, and -3; CAR7-T Cells on day 0.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the primary safety and efficacy of anti-CD7 chimeric antigen receptor(CAR)-modified T cells(CAR7-Ts) in patients with relapsed or refractory T lymphoid malignancies.

DETAILED DESCRIPTION:
Chimeric antigen receptor-T cells (CAR-T) have made breakthroughs in the treatment of B-cell tumors, especially refractory/relapsed acute B lymphocytes. CD7 is a transmembrane glycoprotein expressed by T cells and natural killer cells and their precursors; it is also expressed in >95% of lymphoblastic T-cell leukemias and lymphomas . CD7 was previously evaluated as a target for immunotoxin-loaded antibodies in patients with T-cell malignancies, but tumor responses were limited.

Enhancing the potency of CD7-directed cytotoxicity by substituting donor-derived CAR-T cells for a monoclonal antibody would augment the efficacy of CD7-targeted therapy in patients with T-cell malignancies. To prepare CAR7-T cells, CD7 expression is suppressed on donor-derived T cells by unique blocking technique, and CD7-negative T cells are transduced with a humanized anti-CD7-41BB-CD3ζ lentiviral vector.

This is an investigational study. The objectives are to evaluate the safety and efficacy of CAR7-T cells in patients with CD7+ T-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 14 to 70 years;
2. Expected survival over 60 days;
3. Eastern Cooperative Oncology Group score 0-2;
4. Diagnosed as T-cell hematologic malignancies (including leukemia and lymphoma) according to WHO2016 criteria;
5. Patients must relapse or be refractory after at least two lines of therapy.
6. CD7 were positive in bone marrow or cerebrospinal fluid by immunohistochemistry or flow cytometry at screening, and one of the following conditions is satisfied:

   A. No remission was achieved after at least 2 lines of standard therapy; B. Relapse or progression after standard treatment; C. Relapse after autologous or allogeneic hematopoietic stem cell transplantation;
7. Have no fertility requirements or plans for one year since enrollment in this clinical trial;
8. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.

Exclusion Criteria:

1. Complicated with central system leukemia/lymphoma with active intracranial lesions;
2. Existing or preexisting CNS conditions, such as epileptic seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any CNS related autoimmune disease;
3. Symptomatic heart failure or severe arrhythmias;
4. Symptoms of severe respiratory failure;
5. Complicated with other types of malignant tumors;
6. Serum creatinine and/or urea nitrogen ≥ 1.5 times of normal value;
7. Suffer from sepsis or other uncontrollable infections;
8. Intracranial hypertension or brain consciousness disorder;
9. Severe mental disorders;
10. Have received organ transplantation (excluding bone marrow transplantation);
11. Female patients (fertile patients) had positive blood HCG test;
12. Hepatitis (including hepatitis B and C), AIDS and syphilis were screened positive;
13. Patients with graft-versus-host disease (GVHD) or who require immunosuppressant treatment;
14. The absolute value of lymphocytes was too low to manufacture CART cells;
15. Other conditions considered inappropriate by the researcher.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-04-07 (Estimated); Study Completion 2024-04-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 2 years after infusion
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate(ORR) of administering CAR7-T cells in Relapsed/Refractory CD7+ T-cell hematological malignancies. | within 2 years after infusion
  ORR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Complete response rate(CRR) of administering CAR7-T cells in Relapsed/Refractory CD7+ T-cell hematological malignancies. | within 2 years after infusion
  CRR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Progress-free survival(PFS) of administering CAR7-T cells in Relapsed/Refractory CD7+ T-cell hematological malignancies. | within 2 years after infusion
  PFS will be assessed from CAR T cell infusion to death or last follow-up (censored).
Duration of Response(DOR) of administering CAR7-T cells in Relapsed/Refractory CD7+ T-cell hematological malignancies. | within 2 years after infusion
  DOR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Overall survival(OS) of administering CAR7-T cells in Relapsed/Refractory CD7+ T-cell hematological malignancies. | within 2 years after infusion
  OS will be assessed from CAR T cell infusion to death or last follow-up (censored).

OTHER OUTCOMES:
In vivo expansion and survival of CAR7-T cells | within 2 years after infusion
  Quantity of CAR copies in bone marrow and peripheral blood will be determined by using quantitative polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomes-Silva D, Srinivasan M, Sharma S, Lee CM, Wagner DL, Davis TH, Rouce RH, Bao G, Brenner MK, Mamonkin M. CD7-edited T cells expressing a CD7-specific CAR for the therapy of T-cell malignancies. Blood. 2017 Jul 20;130(3):285-296. doi: 10.1182/blood-2017-01-761320. Epub 2017 May 24. PMID 28539325